CLINICAL TRIAL: NCT00926315
Title: Influence of Vitamin D on Gene Expression Profile of Breast Cancer Samples From Post-menopausal Patients
Brief Title: Gene Expression Profile of Breast Cancer Samples After Vitamin D Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Eduardo Carneiro de Lyra, MD, PhD, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FMUSPIBCCVD2009; CAPPesq 626/06 (Registry Identifier: Comissão Ética para Análise Projetos Pesquisa HCFMUSP 626/06); FAPESP 07/04799-2 (Other Grant/Funding Number: Fundação de Amparo à Pesquisa Estado de São Paulo 07/04799-2); IBCC 108/2006/07 (Registry Identifier: Comitê de Ética em Pesquisa IBCC 108/2006/07); CAPPesq 0018/09 (Registry Identifier: Comissão Ética para Análise Projetos Pesquisa HCFMUSP)
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Breast Neoplasms; Postmenopausal Disorder
Keywords: Breast Neoplasms; Calcitriol; Postmenopausal; Cell Proliferation; Gene Expression Profiling
MeSH Terms: conditions — Breast Neoplasms; Hyperplasia | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- calcitriol (Experimental): calcitriol supplementation (0.25 mcg 2x/d)
  Interventions: Drug: calcitriol

INTERVENTIONS:
Drug: calcitriol — Post menopausal patients will receive Calcitriol 0.50 mcg PO per day for 1 month.
  Other Names: Rocaltrol
Drug: Calcitriol — calcitriol 0.25 mcg PO bid
  Other Names: Rocaltrol

SUMMARY:
The purpose of this study is to evaluate whether calcitriol supplementation may reduce tumor cell proliferation and influence gene expression profile of breast cancer samples from post-menopausal patients.

DETAILED DESCRIPTION:
Women affected by breast cancer present lower 1,25(OH)2D3 or 25(OH)D3 serum levels than unaffected ones. Calcitriol supplementation may be indicated to post-menopausal women to reduce bone loss. Vitamin D has antiproliferative effects in breast cancer cell lines and breast cancer xenografts.

Post-menopausal breast cancer patients will be prescribed calcitriol supplementation, in doses indicated to prevent osteoporosis, while they are submitted to biopsy, staging exams and have their breast surgery scheduled (approximately one month). Tumor dimension and proliferation rate (as determined by Ki67 expression), 25(OH)D3 and/or 1,25(OH)2D3 serum concentration, will be evaluated before and after calcitriol supplementation. Tumor gene expression will be evaluated in samples collected before and after supplementation to analyze the differential profile.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Invasive breast carcinoma
* Clinical conditions for breast surgery
* No previous neoadjuvant treatment for breast cancer
* Agreement to take part in the study and sign the informed consent

Exclusion Criteria:

* History of hypercalcemia or nephrolithiasis
* Current use of corticosteroids, vitamin D supplementation, HRT
* Previous chemotherapy, hormonotherapy or radiotherapy
* Parathyroid disease
* Absence of clinical condition to receive supplementation

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Tumor dimension and proliferation evaluated by ultrasound and Ki67 expression; Tumor gene expression profile | 30 days

SECONDARY OUTCOMES:
Follow-up for 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Aparecida A Koike Folgueira, MD,PhD, Study Chair — Faculdade de Medicina - Universidade de São Paulo; Eduardo Carneiro de Lyra, MD, PhD, Principal Investigator — Instituto Brasileiro de Controle do Cancer; Yuri N Urata, MSc, Principal Investigator — Faculdade de Medicina da Universidade de São Paulo; Maria Lucia H Katayama, PhD, Principal Investigator — Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] de Lyra EC, da Silva IA, Katayama ML, Brentani MM, Nonogaki S, Goes JC, Folgueira MA. 25(OH)D3 and 1,25(OH)2D3 serum concentration and breast tissue expression of 1alpha-hydroxylase, 24-hydroxylase and Vitamin D receptor in women with and without breast cancer. J Steroid Biochem Mol Biol. 2006 Aug;100(4-5):184-92. doi: 10.1016/j.jsbmb.2006.04.009. Epub 2006 Jul 7. PMID 16828283
- [Background] Rozenchan PB, Folgueira MA, Katayama ML, Snitcovsky IM, Brentani MM. Ras activation is associated with vitamin D receptor mRNA instability in HC11 mammary cells. J Steroid Biochem Mol Biol. 2004 Sep;92(1-2):89-95. doi: 10.1016/j.jsbmb.2004.05.007. PMID 15544934
- [Background] Katayama ML, Pasini FS, Folgueira MA, Snitcovsky IM, Brentani MM. Molecular targets of 1,25(OH)2D3 in HC11 normal mouse mammary cell line. J Steroid Biochem Mol Biol. 2003 Jan;84(1):57-69. doi: 10.1016/s0960-0760(03)00004-9. PMID 12648525
- [Background] Bortman P, Folgueira MA, Katayama ML, Snitcovsky IM, Brentani MM. Antiproliferative effects of 1,25-dihydroxyvitamin D3 on breast cells: a mini review. Braz J Med Biol Res. 2002 Jan;35(1):1-9. doi: 10.1590/s0100-879x2002000100001. PMID 11743608
- [Background] Folgueira MA, Federico MH, Katayama ML, Silva MR, Brentani MM. Expression of vitamin D receptor (VDR) in HL-60 cells is differentially regulated during the process of differentiation induced by phorbol ester, retinoic acid or interferon-gamma. J Steroid Biochem Mol Biol. 1998 Aug;66(4):193-201. doi: 10.1016/s0960-0760(98)00041-7. PMID 9744516
- [Background] Janjoppi L, Katayama MH, Scorza FA, Folgueira MA, Brentani M, Pansani AP, Cavalheiro EA, Arida RM. Expression of vitamin D receptor mRNA in the hippocampal formation of rats submitted to a model of temporal lobe epilepsy induced by pilocarpine. Brain Res Bull. 2008 Jul 30;76(5):480-4. doi: 10.1016/j.brainresbull.2008.01.002. Epub 2008 Feb 5. PMID 18534255
- [Background] Folgueira MA, Carraro DM, Brentani H, Patrao DF, Barbosa EM, Netto MM, Caldeira JR, Katayama ML, Soares FA, Oliveira CT, Reis LF, Kaiano JH, Camargo LP, Vencio RZ, Snitcovsky IM, Makdissi FB, e Silva PJ, Goes JC, Brentani MM. Gene expression profile associated with response to doxorubicin-based therapy in breast cancer. Clin Cancer Res. 2005 Oct 15;11(20):7434-43. doi: 10.1158/1078-0432.CCR-04-0548. PMID 16243817